CLINICAL TRIAL: NCT05782348
Title: Clinical Study to Evaluate the Effectiveness of a Cognitive Behavioral Intervention (CBI) Adjunctive to a Smart Powered Toothbrush on the Oral Health of Adolescents
Brief Title: Evaluating the Effectiveness of a Cognitive Behavioral Intervention (CBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Howard University (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Brian Laurence, Professor, Howard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRO-2022-10-CBT-HU-US-BS
Record Dates: First submitted 2023-03-02; First posted 2023-03-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Adolescent Behavior; Dental Plaque; Gingivitis; Cognitive Change
Keywords: adolescent health; dental plaque; gingivitis; cognitive change
MeSH Terms: conditions — Adolescent Behavior; Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: Three arm parallel group single blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Group I (Experimental): A commercially available fluoride toothpaste (1450 ppm F) A commercially available Smart Electric toothbrush Cognitive behavioral intervention (CBI)
  Interventions: Behavioral: Cognitive behavioral intervention; Other: Colgate smart toothbrush
- Control group I (Active Comparator): A commercially available fluoride toothpaste (1450 ppm F) A commercially available Smart Electric toothbrush
  Interventions: Other: Colgate smart toothbrush
- Control group II (No Intervention): A commercially available fluoride toothpaste (1450 ppm F) A commercially available soft bristle toothbrush

INTERVENTIONS:
Behavioral: Cognitive behavioral intervention — A six-session CBI Intervention component will be used with the TEST GROUP I. This will examine a cognitive behavioral intervention designed to improve tooth brushing and oral hygiene. The components include oral health education, values-based activities, motivational interviewing, goal setting, problem solving skills, cognitive restructuring, verbal reinforcement and stress management.
  Arms: Test Group I
Other: Colgate smart toothbrush — A Colgate smart toothbrush that provides the user with details on toothbrushing habits and frequency
  Arms: Control group I; Test Group I

SUMMARY:
This is a Phase III, randomized, one-center, three arm parallel group, open label and single blind clinical study to evaluate the effectiveness of a cognitive behavioral intervention (CBI) adjunctive to a smart powered toothbrush on the oral health of adolescents.

DETAILED DESCRIPTION:
This is a Phase III, randomized, one-center, three arm parallel group, open label and single blind clinical study to evaluate the effectiveness of a cognitive behavioral intervention (CBI) adjunctive to a smart powered toothbrush on the oral health of adolescents. Outcomes briefly summarized include the plaque score, gingival score and a survey of knowledge, attitudes and procedures measured at 1,3 and 6 months

Participating subjects will be randomized to one of the following products:

TEST GROUP I A commercially available fluoride toothpaste (1450 ppm F) A commercially available Smart Electric toothbrush CONTROL GROUP I A commercially available fluoride toothpaste (1450 ppm F) A commercially available Smart Electric toothbrush CONTROL GROUP II A commercially available fluoride toothpaste (1450 ppm F) A commercially available soft bristle toothbrush

ELIGIBILITY:
Inclusion Criteria:

Students are enrolled in participating high schools Caregivers give informed consent Student gives assent

Exclusion Criteria:

* Having a prosthetic heart valve
* Having a history of previously having infective endocarditis
* Having had joint replacement surgery
* Children on blood thinner medication such as Coumadin or Rivaroxaban
* Children who are currently receiving chemotherapy
* Children who have received organ transplants of any type
* Children with Leukemia

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2023-08-06 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Gingival inflammation | All outcomes will be measured at baseline, at1 month, 3 months and at 6 months
  A Löe-Silness Gingival Index score from 0 to 3 will be assigned by the examining dentist to all scorable surfaces of the maxillary and mandibular teeth using a dental light and dental mirror. A whole mouth mean score for each subject will be determined by adding the values given by the examining dentist to each scorable surface and dividing that number by the total number of surfaces scored.
  Scores Criteria 0 Absence of inflammation
  1. Mild inflammation- Slight change in color and mild edema with little change in texture. No bleeding on probing.
  2. Moderate inflammation- moderate glazing, redness, edema and hypertrophy. Bleeding on probing.
  3. Severe inflammation- Marked redness, hypertrophy, edema and ulceration. Tendency for spontaneous bleeding.

SECONDARY OUTCOMES:
Plaque scores | All outcomes will be measured at baseline, 1 month, 3 months and at 6 months
  Mean plaque index scores will be computed for each subject. Each tooth is scored in six areas: 1) mesio-facial; 2) mid-facial; 3) disto-facial; 4) mesio-lingual; 5) mid-lingual; and 6) disto-lingual. Whole mouth within subject mean scores will be computed as follows:
  Total plaque score for all scoring sites divided by total number of scoring sites
Knowledge assessment | All outcomes will be measured at baseline, 1 month, 3 months and at 6 months
  Knowledge will be assessed using 19 item scale previously used by the researchers
  Enrolled subjects will complete a questionnaire on oral health knowledge, attitudes, and practices including: frequency of brushing and flossing, knowledge, oral health values scale, self-efficacy and motivation. The outcome will be assessed using a 19-item multiple choice survey previously used in Colgate-sponsored research protocols. A six-item oral health self-efficacy scale will be used to measure participant self-reported confidence in their ability to carry out an oral health care routine. Lastly, motivation to engage in recommended oral hygiene behavior will be assessed with a single item 1analog scale (i.e., "How important is it to follow guidelines for brushing twice per day and flossing once per day, from 0 "not important at all" to 10 "most important.")
Efficacy assessment | All outcomes will be measured at baseline, 1 month, 3months and at 6 months
  Efficacy will be assessed using a validated 6 item oral health self-efficacy scale
Motivation assessment | All outcomes will be measured at baseline, 1 month, 3months and at 6 months
  Motivation will be assessed using a single item 10-point visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Friendship Public Charter School, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available to other researchers